CLINICAL TRIAL: NCT00079443
Title: A Phase II Study of Single Agent Depsipeptide (NSC 630176) Followed by a Phase I Study of Rituximab/Fludarabine Combination With an Escalating Dose of Depsipeptide in Relapsed or Refractory Low Grade B Cell Lymphomas
Brief Title: FR901228 Alone or Combined With Rituximab and Fludarabine in Treating Patients With Relapsed or Refractory Low-Grade B-Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00043; UMGCC #0307; MSGCC-0307; CDR0000355763; NCI-6015; U01CA069854 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — romidepsin; Rituximab; fludarabine phosphate

ARMS (1):
- Treatment (Experimental): PHASE II: Patients receive FR901228 IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Patients who achieve a complete or partial remission receive 2 additional courses (for a total of 6 courses). Patients with stable disease after 4 courses or progressive disease at any time after 2 courses proceed to the phase I portion of the study.
  PHASE I: Patients receive rituximab IV over approximately 4-8 hours on day 1; fludarabine IV over 10-30 minutes on days 2-4; and FR901228 IV over 4 hours on days 2, 9, and 16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin; Biological: rituximab; Drug: fludarabine phosphate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the best dose of FR901228 when given together with rituximab and fludarabine and to see how well FR901228 works alone in treating patients with relapsed or refractory low-grade B-cell non-Hodgkin's lymphoma. Drugs used in chemotherapy, such as FR901228 and fludarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Rituximab may increase the effectiveness of chemotherapy drugs by making cancer cells more sensitive to the drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. For phase 2: is to assess the clinical efficacy (complete and partial response rates) of single agent depsipeptide.

II. For phase 1: is to assess the feasibility of adding Depsipeptide to a regimen of Rituximab and Fludarabine and to establish the MTD of Depsipeptide in this combination.

SECONDARY OBJECTIVES:

I. To correlate disease response (clinical outcome) with the changes in histone acetylation assays.

II. Study the expression of death receptors of DR4 and DR5 after treatment with depsipeptide.

III. Assessment of minimal residual disease by immune histochemistry.

OUTLINE: This is a multicenter, phase II study of single-agent FR901228 followed by a phase I, dose-escalation study of FR901228.

PHASE II: Patients receive FR901228 IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients who achieve a complete or partial remission receive 2 additional courses (for a total of 6 courses). Patients with stable disease after 4 courses or progressive disease at any time after 2 courses proceed to the phase I portion of the study.

PHASE I: Patients receive rituximab IV over approximately 4-8 hours on day 1; fludarabine IV over 10-30 minutes on days 2-4; and FR901228 IV over 4 hours on days 2, 9, and 16. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of FR901228 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for up to 3 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and clinically confirmed relapsed and/or refractory low grade follicular B cell NHL (follicular small cleaved cell, follicular mixed small and large cell, and small lymphocytic lymphoma (according to the IWF classification); the malignant tissues must be positive for CD 20 on immunohistochemistry or flow cytometry
* History of one or multiple prior chemotherapy regimens for low grade follicular NHL, but no more than 4 therapies

  * For the phase II trial: previous therapies can include rituximab, fludarabine (alone not in combination or sequentially); the most recent therapy should be completed more then 4 weeks prior to protocol entry, 6 months if the last regimen included Fludarabine, rituximab, nitrosoureas or mitomycin, and at least 8 weeks out from a treatment with UCN-01
  * For phase I trial: Patients can move from phase II to phase I trial if they have not received rituximab and fludarabine in combination or sequentially in the past, if they received one or both agents individually and had a 50% responses; this response corresponds to PR to prior therapy
* Presence of measurable disease by CT scan 4 weeks after the last chemotherapeutic regimen with at least one lesion greater than 1.5c m in one dimension and or positive bone marrow biopsy
* ECOG performance status ≤ 2 with a minimal life expectancy of 4 months
* Female patients of childbearing age should have negative pregnancy test; pregnant and breast-feeding women will not be eligible for the study because the antiproliferative effects of depsipeptide may be harmful to the developing fetus or nursing infants
* Absolute neutrophil count >= 1000/µl; lower ANC (>= 500/µl) count will be considered if they are due to a bone marrow involvement by the disease; patients can receive growth factors (G-CSF and erythropoietin) to sustain the peripheral counts during the cycles of therapy
* Platelets >= 100.000/µl; lower platelets (>50.000/µl) count will be considered if they are due to a bone marrow involvement by the disease; patients can receive growth factors (G-CSF and erythropoietin) to sustain the peripheral counts during the cycles of therapy
* Total bilirubin =< 1.5 x institutional upper limit of normal
* AST/ALT =< 3 x institutional upper limit of normal
* Creatinine =< 1.5 x the institutional upper limit of normal
* Patients with history of seizures are included if under adequate control; blood levels of seizure medications are monitored during the study
* The patient must understand the investigational nature of the protocol, potential risks and benefits of the study and provides an informed written consent form

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (within 6 weeks for rituximab, nitrosoureas and mitomycin and within 8 weeks for UCN-01) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who had prior treatment with depsipeptide or any other histone deacetylase inhibitor
* Patients who had prior allogeneic stem cell transplantation
* Bulky disease: single mass greater than or equal to 10 cm
* Patients may not be receiving any other investigational agents
* Patients with known CNS involvement (as documented by MRI and or cerebro-spinal fluid examination) should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events
* History of life threatening allergic reactions attributed to agents used in the study
* Impaired cardiac function: history of life threatening arrhythmias, MI within the preceding 6 months, severe CAD, cardiomyopathy, congestive heart failure >= NYH II; EF =< 40%; EKG abnormality i.e.: ischemic ST-T abnormalities, QT prolongation, pathologic q waves, arrhythmias (except for benign PAC's and PVC's, 1st degree AV block, 2nd degree AV block Wenkebach); patients with LVH on EKG will be ineligible for this trial
* Patients with prior malignancies other then basal cell carcinomas and cervical intra-epithelial neoplasia
* Patients (or their partners) unwilling to use contraception
* Patients who require pharmacological doses of corticosteroids for intercurrent medical conditions
* Patients who uses concomitant drugs which may cause a prolongation of QTc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-01; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (Phase II) | Up to 3 years
  Exact confidence interval of the response rate will be calculated.
Survival (Phase II) | Up to 3 years
  Kaplan-Meier analysis will be used to describe patient survival.
MTD, defined as the highest dose level at which 6 patients have been treated with not more than 1 DLT, graded according to NCI CTC version 2 (Phase I) | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Badros, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States